CLINICAL TRIAL: NCT02768571
Title: Effects of Cerebrolysin Combined With Rehabilitation on Motor Recovery in Patients With Severe Motor Involvement at Subacute Phase of Stroke
Brief Title: Effects of Cerebrolysin Combined With Rehabilitation on Motor Recovery in Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Ever Neuro Pharma GmbH (Industry)
Responsible Party: Principal Investigator, Yun-Hee Kim, Professor, MD, PhD, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-10-034
Record Dates: First submitted 2016-03-04; First posted 2016-05-11 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Stroke
Keywords: cerebrolysin, stroke, motor function
MeSH Terms: conditions — Stroke | interventions — cerebrolysin; brain natriuretic peptide, porcine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cerebrolysin (Experimental): Cerebrolysin 30 ml with 100 ml dilution/day * 21 days with rehabilitation
  * Study drug schedule - given from day 8 after stroke, but, if day 8 is weekend, the given day is the next Monday(day 9~10)
  * Rehabilitation
    * 3 hours (physiotherapy: 2 hours, occupational therapy: 1 hour) / day
    * 5 times/week for 3 weeks
  Duration of Treatment:
  Study drug will be given once daily by intravenous infusion for 21 consecutive days on study day 8 ~ 28.
  The clinical observation period for each patient will be 90 days and will include four clinical evaluation visits at Screening(day ≤ 7), Baseline(day 8) and on study day 29, and 90.
  Interventions: Drug: Cerebrolysin
- Placebo (Placebo Comparator): Saline 100 ml/day * 21 days with rehabilitation
  * Study drug schedule - given from day 8 after stroke, but, if day 8 is weekend, the given day is the next Monday(day 9~10)
  * Rehabilitation
    * 3 hours (physiotherapy: 2 hours, occupational therapy: 1 hour) / day
    * 5 times/week for 3 weeks
  Duration of Treatment:
  Study drug will be given once daily by intravenous infusion for 21 consecutive days on study day 8 ~ 28.
  The clinical observation period for each patient will be 90 days and will include four clinical evaluation visits at Screening(day ≤ 7), Baseline(day 8) and on study day 29, and 90.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cerebrolysin — Cerebrolysin- cerebrolysin 30 ml with 100 ml dilution/day * 21 days with rehabilitation
  Other Names: Porcine brain peptide
  Arms: Cerebrolysin
Drug: Placebo — Placebo- saline 100 ml/day * 21 days with rehabilitation
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This study, E-COMPASSII is a phase IV clinical trial designed as a multicenter, randomized, double-blind, placebo-controlled, parallel-group study. This study will enroll 80 subacute stroke patients with severe motor involvement. Primary objective is to demonstrate the efficacy of porcine brain peptide to improve motor recovery measured by the improvement ratio of Fugl-Meyer assessment ((score of FMA after 3 weeks - score of FMA at baseline) / score of FMA at baseline) in patients with subacute stroke. Secondary objectives are to evaluate the safety profile of cerebrolysin and to test the hypothesis that subacute stroke patients with severe motor involvement randomized to administration of Cerebrolysin combined with rehabilitation for 3 weeks show better outcome on global function (Korean version Modified Barthel Index, K-MBI), severity of stroke (National Institute of Health Stroke Scale, NIHSS), cognitive function (Korean Version of Mini-Mental State Exam, K-MMSE; Korean version Montreal Cognitive Assessment, K-MoCA), upper limb function (Action Research Arm Test, ARAT; Box and block test, B&B) and neuroplasticity measure (resting-state functional MRI(rsfMRI), diffusion tensor image(DTI), and motor evoked potential(MEP)) at 3 months after stroke.

DETAILED DESCRIPTION:
Randomized double-blinded, placebo-controlled multicenter study with two treatment groups

Number of Patients: 80 patients (n = 40 per group) 5 study centers will participate in this study.

Group 1(Cerebrolysin): cerebrolysin 30 ml with 100 ml dilution/day * 21 days with rehabilitation

Group 2(Placebo): saline 100 ml/day * 21 days with rehabilitation

ELIGIBILITY:
Inclusion Criteria:

1. The first-ever stroke (ischemic)
2. Confirmed by CT or MRI
3. Subacute stage: less than 1 week
4. Severe motor function involvement (FMA < 50)
5. Age: between 19 and 80 years
6. Inpatients
7. Written informed consent obtained from the patient or legally authorized representative

Exclusion Criteria:

1. Contraindication of MRI
2. Progressive or unstable stroke
3. Pre-existing and active major neurological disease
4. Pre-existing and active (e.g., on chronic medication) major psychiatric disease, such as major depression, schizophrenia, bipolar disease, or dementia
5. A history of significant alcohol or drug abuse in the prior 3 years
6. Advanced liver, kidney, cardiac, or pulmonary disease
7. A terminal medical diagnosis consistent with survival < 1 year
8. Substantial decrease in alertness at the time of randomization, defined as score of 2 on NIH Stroke Scale
9. Pregnancy or lactating; note that a negative pregnancy test will be required if the patient is a female in reproductive years
10. Any condition that would represent a contraindication to Cerebrolysin, including allergy to Cerebrolysin
11. Current enrolment in another therapeutic study of stroke or stroke recovery
12. Total serum bilirubin > 4 mg/dL, alkaline phosphatase > 250 U/L, SGOT/AST > 150 U/L, SGPT/ALT > 150 U/L, or creatinine > 3.5 mg/dL; or cardiopulmonary deficits large enough to interfere with reasonable participation in physiotherapy during the trial.
13. Previous porcine brain peptide administration history

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Score of Fugl-Meyer assessment (FMA) | 3 months after stroke
  Motor function

SECONDARY OUTCOMES:
Score of Korean version Modified Barthel Index (K-MBI) | 3 months after stroke
  Global function
Score of National Institute of Health Stroke Scale (NIHSS) | 3 months after stroke
  Severity of stroke
Score of Korean Version of Mini-Mental State Exam(K-MMSE) and Korean version of Montreal Cognitive Assessment (K-MoCA) | 3 months after stroke
  Cognitive function
Score of Action Research Arm Test (ARAT) and box and block test | 3 months after stroke
  Upper limb function
Score of EuroQol (EQ-5D) | 3 months after stroke
  Quality of life
Days of Length of hospital stay | 3 months after stroke
Brain activation of resting-state functional MRI | 3 months after stroke
  Neuroplasticity measure

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, MD, PhD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No